CLINICAL TRIAL: NCT02811198
Title: Pain, Reward, Attention and Neurocircuitry: Biomarkers of Suicidality
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: SBIO-01
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder; Suicide; Suicidal Ideation
MeSH Terms: conditions — Depressive Disorder, Major; Suicide; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for genetic and proteomic analysis. Saliva samples will be collected to measure cortisol levels.

GROUPS / COHORTS (4):
- MDD with SI and No Attempt: Subjects will have MDD with current MDE, current suicidal ideation and no lifetime suicide attempts
  Interventions: Other: No intervention
- MDD with SI and Recent Attempt: Subjects with have MDD with current MDE, current suicidal ideation and a suicide attempt within the past 6 months
  Interventions: Other: No intervention
- MDD with no SI and Lifetime Attempt: Subjects with MDD and current MDE but no current suicidal ideation and a lifetime suicide attempt.
  Interventions: Other: No intervention
- Healthy Controls: Subjects will have no personal or family psychiatric history and no suicide attempts.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The ultimate aim of this study is to identify a biomarker of suicide risk in MDD by measuring the "hedonic spectrum" (pain and reward responsivity), attention and its associated brain structures using brain scans (fMRI and DTI), as well as the stability of markers over time.

DETAILED DESCRIPTION:
The issue of suicide has continued to puzzle researchers in the field of psychiatry. Edwin Shneidman, a prominent researcher on suicide emphasized "the most evident fact about suicidology and suicidal events is that they are multidimensional…containing concomitant biological, sociological, and psychological (interpersonal and intrapsychic)…elements". Yet, no study to date has attempted to integrate these dimensions when evaluating suicide risk. Considering the presence of a psychiatric illness is a primary predictor of suicide, it is important to develop a unified understanding of risk factors that integrate current clinical and neurobiological findings in this population.

Our aim is to: (1) identify an integrated biomarker model to predict risk of suicide attempt in patients with Major Depressive Disorder (MDD) with and without a history of suicide attempt, using neuroimaging, neurocognitive testing and behavioural tasks, and (2) test the stability of this model using a prospective 1 year design.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 criteria for Major Depressive Episode within a MDD, confirmed through MINI diagnosis104
2. Ages between 18 and 70 years
3. Hamilton Depression Rating Scale - 17 item (HAMD-17) >= 14
4. Capable of giving informed consent
5. Groups 1 and 2 participants only: HAMD-17 item 3 (suicide) >= 2
6. Group 2 participants only: positive history of a suicide attempt within the last six months
7. Group 3 participants only: positive history of a lifetime suicide attempt

Exclusion Criteria:

1. Pregnancy/lactation
2. Medical condition requiring immediate investigation or treatment
3. Recent (< 6 months)/current history of drug abuse/dependence (other than caffeine, or nicotine)
4. Lifetime history of psychosis, Bipolar I or Bipolar II; other Axis I comorbidities are allowable
5. Individuals who are taking a daily sedative hypnotic, atypical antipsychotic or stimulant must be on a stable dose for at least 4 weeks prior to the neuroimaging scan. The dose must not be taken after 10:00pm the evening prior to the scan. Those receiving a benzodiazepine or an atypical antipsychotic on an "as needed" basis (taken, but not every day) will be washed out of their benzodiazepine/atypical antipsychotic for two weeks prior to neuroimaging. Those receive stimulants on an "as needed" basis will be washed out for 1-3 days prior to neuroimaging, depending on the stimulant half-life.
6. Participation in experimental treatment trials for the study duration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will recruited from Mental Health Clinics at St. Michael's Hospital from Mood Disorders Clinics, University Health Networks (UHN) hospitals, and self-referrals from advertisements in Mental Health Department, and on social media.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Biomarkers for Suicide Risk | 12 months
  Potential biomarkers for suicide risk including brain scans, genomic or proteomic makers,

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Sakina Rizvi, Toronto, Ontario, Canada